CLINICAL TRIAL: NCT03882775
Title: Bivalirudin vs Heparin in Elderly Patients With Acute ST-segment Elevation Myocardial Infarction Undergoing Emergency Percutaneous Coronary Intervention
Brief Title: Bivalirudin in Elderly Patients With Acute ST-segment Elevation Myocardial Infarction
Acronym: BEST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PJ-KY-2018-117
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: STEMI; Percutaneous Coronary Intervention; Aged
Keywords: Major adverse cardiac events (MACEs); bivalirudin
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Cardiovascular Diseases | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bivalirudin (Experimental): Bivalirudin will be given as a bolus of 0.75 mg/kg followed by infusion of 1.75 mg/kg/h during the PCI procedure and for at least 30 minutes but no more than 4 hours afterwards. Following this mandatory infusion,a reduced-dose infusion (0.2 mg/kg/h) for up to 20 hours could be administered at physician discretion. An additional bivalirudin bolus of 0.3 mg/kg was given if the activated clotting time 5 minutes after the initial bolus was less than 225 seconds.
  Interventions: Drug: Bivalirudin
- Heparin (Active Comparator): Heparin will be administered at a dose of 70 to 100 units per kilogram in patients not receiving glycoprotein IIb/IIIa inhibitors and at a dose of 50 to 70 units per kilogram in patients receiving glycoprotein IIb/IIIa inhibitors. Subsequent adjustment of the heparin dose on the basis of the activated clotting time will be left to the discretion of the treating physicians.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin — Patients would be given anticoagulant therapy with bivalirudin in acute STEMI during emergency PCI operation.
  Arms: Bivalirudin
Drug: Heparin — heparin with or without gpi during emergency PCI.
  Arms: Heparin

SUMMARY:
The study is an investigator-sponsored, prospective, multicenter, randomized, open-label study designed to compare efficacy and safety between bivalirudin and heparin in elderly patients with acute ST-segment elevation myocardial infarction undergoing emergency PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥75 years old;
* Planned emergency (Symptom onset within 24h) PCI for acute STEMI patients;
* Life expectancy ≥ 1 year;
* Provide written informed consent.

Exclusion Criteria:

* Contraindications to angiography or PCI;
* Active bleeding or bleeding constitution, bleeding tendency, including GI or urinary tract hemorrhage (3 months), cerebral hemorrhage (6 months) or cerebral infarction history (3 months), etc;
* Other disease may lead to vascular lesions and secondary bleeding factors (such as active gastric ulcer, active ulcerative colitis, intra-cerebral mass, aneurysm, etc.);
* Severe renal insufficiency (eGFR < 30 mL/min/ 1.73 m2);
* Elevated AST, ALT level higher than three times of the normal upper limit;
* Advanced heart failure (NYHA classification grading of cardiac function ≥ Ⅲ)
* Complicated with immune system diseases；
* Abnormal hematopoietic system：platelet count < 100 * 109 / L or > 700 * 109 / L，white blood cell count < 3 * 109/L etc;
* Suffering from acute infections ,infectious diseases or other serious diseases, such as malignant tumors;
* Known intolerance, or contraindication to any antithrombotic medication
* Known allergy to the study drugs and instruments (UFH, bivalirudin, aspirin and clopidogrel, stainless steel, contrast agents, etc.), or those allergic constitution.
* Non-cardiac co-morbid conditions are present that may result in protocol non-compliance;
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period;
* Patient's inability to fully cooperate with the study protocol

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-07-14 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 7 days
  a composite of cardiac death, reinfarction, heart failure,ischemic stroke,frequent post infarction angina，Ventricular tachycardia or fibrillation requiring electrical cardioversion or defibrillation.
Major bleeding | 7 days
  BARC types 3-5 bleeding;TIMI major bleeding or GUSTO moderate to severe bleeding

SECONDARY OUTCOMES:
Major adverse cardiac events | 30 days
  a composite of cardiac death, reinfarction, heart failure,ischemic stroke,frequent post infarction angina，Ventricular tachycardia or fibrillation requiring electrical cardioversion or defibrillation.
Stent thrombosis ,TVR ,TLR | 30 days
  rate of stent thrombosis,unplanned target-vessel revascularization and target lesion revascularisation
Major adverse cardiac events | 180 days
  a composite of cardiac death, reinfarction, heart failure,ischemic stroke,frequent post infarction angina，Ventricular tachycardia or fibrillation requiring electrical cardioversion or defibrillation.
Stent thrombosis ,TVR ,TLR | 180 days
  rate of stent thrombosis,unplanned target-vessel revascularization and target lesion revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Rongchong Huang, M.D., Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

REFERENCES:
- [Background] De Caterina R, Husted S, Wallentin L, Andreotti F, Arnesen H, Bachmann F, Baigent C, Huber K, Jespersen J, Kristensen SD, Lip GY, Morais J, Rasmussen LH, Siegbahn A, Verheugt FW, Weitz JI; European Society of Cardiology Working Group on Thrombosis Task Force on Anticoagulants in Heart Disease. Parenteral anticoagulants in heart disease: current status and perspectives (Section II). Position paper of the ESC Working Group on Thrombosis-Task Force on Anticoagulants in Heart Disease. Thromb Haemost. 2013 May;109(5):769-86. doi: 10.1160/TH12-06-0403. Epub 2013 Mar 28. PMID 23636477
- [Background] Hirsh J, Anand SS, Halperin JL, Fuster V; American Heart Association. AHA Scientific Statement: Guide to anticoagulant therapy: heparin: a statement for healthcare professionals from the American Heart Association. Arterioscler Thromb Vasc Biol. 2001 Jul;21(7):E9-9. doi: 10.1161/hq0701.093520. No abstract available. PMID 11451763
- [Background] Robson R, White H, Aylward P, Frampton C. Bivalirudin pharmacokinetics and pharmacodynamics: effect of renal function, dose, and gender. Clin Pharmacol Ther. 2002 Jun;71(6):433-9. doi: 10.1067/mcp.2002.124522. PMID 12087346